CLINICAL TRIAL: NCT01174771
Title: Noninvasive Cortical Stimulation (rTMS) for Motor and Non-Motor Features of Progressive Supranuclear Palsy (PSP) and Corticobasal Degeneration (CBD)
Brief Title: Repetitive Transcranial Magnetic Stimulation (TMS) for Progressive Supranuclear Palsy and Corticobasal Degeneration
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Choi Deblieck, PhD, University of California, Los Angeles
Other Study IDs: UCaliforniaLA; CurePSP (Other Grant/Funding Number: CurePSP)
Record Dates: First submitted 2010-07-28; First posted 2010-08-04 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Degeneration; Parkinsonism
Keywords: Transcranial magnetic stimulation; Cortical excitability; parkinsonism; Progressive Supranuclear Palsy; Corticobasal Degeneration; PSP; CBD; CBGD
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PSP patients: People that have been clinically diagnosed with atypical parkinsonism, i.e., PSP
- CBD patients: People that have been clinically diagnosed with atypical parkinsonism, i.e., CBD
- Age-matched healthy controls: People that have not been diagnosed with any kind of neurologic movement disorder.

SUMMARY:
Drug therapy of atypical parkinsonism is generally considered either ineffective or minimal 1. Therefore, there is an urgent need to find alternative therapies to treat atypical parkinsonian disorders. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive tool that modulates cortical excitability with minimal discomfort and holds therapeutic promise in treating neurological and psychiatric disorders.

The basal ganglia-thalamocortical circuits that are affected in Progressive Supranuclear Palsy (PSP) and Corticocbasal Ganglionic Degeneration (CBGD) are likely structurally and functionally segregated. The 'motor' circuit is implicated in parkinsonian akinesia and hypokinesia; a 'prefrontal' circuit is implicated in working memory and mood regulation, and linked with non-motor symptoms such as depression and apathy. In this proposal, we characterize motor and prefrontal network dysfunction in PSP and CBGD patients, and propose that high-frequency and low-frequency rTMS directed over separate motor and prefrontal cortical targets of each network may show specific and selective beneficial effects on motor vs. cognitive function in PSP and CBGD patients, respectively. Quantitative motor outcome measures include timed finger tapping tasks. Quantitative cognitive outcome measures comprise a visual analogue scale (VAS).

If successful, this pilot study will provide proof of principle data to suggest potential benefits for rTMS in PSP/CBGD patients, and provide sufficient data and experience to support future PSP/CBGD studies that include the use of rTMS to investigate the pathophysiology of motor and non-motor features of PSP and CBGD patients.

DETAILED DESCRIPTION:
Background: Drug therapy of atypical parkinsonism is generally ineffective or minimal, and novel therapy approaches for atypical parkinsonian disorders are needed. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive tool that modulates cortical excitability and holds promise in treating neurological/psychiatric disorders. The 'motor' basal ganglia-cortical circuit is implicated in parkinsonian akinesia and hypokinesia; a 'prefrontal' circuit is implicated in working memory (WM) and mood regulation, possibly linked to depression and apathy.

Hypothesis: Motor deficits in Progressive Supranuclear Palsy (PSP) and Corticobasal Ganglionic Degeneration (CBGD) are associated with a dysfunctional motor network; emotional deficits in PSP/CBGD are associated with a dysfunctional prefrontal network. We hypothesize that high-frequency and low-frequency rTMS over cortical targets will selectively and specifically improve tasks and symptoms relevant to that target in PSP and CBGD patients, respectively.

Aims: To contrast cortical excitability characteristics and motor and emotional function between PSP and CBGD patients. To determine selective and specific beneficial rTMS effects over primary motor (M1) and dorsolateral prefrontal (DLPFC) cortex on cortical excitability characteristics and motor and emotional function in PSP and CBGD patients.

Design: Ten individuals with PSP and ten with CBGD will participate in a within-subject cross-sectional design. Motor outcome measures include a timed finger tapping task at comfortable and maximal speed. Quantitative cognitive outcome measures comprise a visual analogue scale of mood states (VAS). After a first baseline visit, PSP patients will receive high-frequency 5 Hz rTMS in two separate visits to two site conditions (left DLPFC vs. the more affected side of M1) across subjects with two within-session task conditions (motor vs. cognitive). They will also receive sham stimulation in a separate visit. These three stimulation visits will be randomized. CBGD patients will receive the same treatment with the only difference that they will receive low-frequency 1 Hz rTMS instead.

Relevance: If successful, we will demonstrate a double-dissociation and causal functional significance between rTMS modulation of M1 in motor tasks and DLPFC in emotional function in PSP Vs. CBGD. Exploratory aims will be conducted. Sufficient data and experience for future PSP/CBGD intervention studies will help identify candidate TMS parameters that are optimal for given symptoms.

ELIGIBILITY:
Inclusion Criteria:

If you are an adult with PSP or CBGD:

1. Must be in good physical health.

If you are neurologically healthy volunteers:

1. Must be older than 35 years

Exclusion Criteria:

1. Must have no implanted metal. Dental fillings are acceptable.
2. Must have no personal seizure or 1st degree relative with history of seizures
3. Must not take any medication that lowers seizure threshold.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The purpose of this study is to learn more about how transcranial magnetic stimulation (TMS) affects motor and non-motor function in patients with Progressive Supranuclear Palsy (PSP) or Cortical Basal Ganglionic Degeneration (CBGD)-forms of parkinsonism.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cortical excitability (CE) measures expressed in motor evoked potentials (MEP) | 1 hour
  We assess cortical excitability (CE) with motor evoked potentials (MEP) and cortical silent periods (CSP) before and after repetitive Transcranial Magnetic Stimulation (TMS).

SECONDARY OUTCOMES:
visual analog scale (VAS) | 2 min
  We assess mood with a visual analog scale (VAS) of 5 emotions and 1 overall feeling of well-being.
tapping speed | 5 min
  tapping speed (movement time and reaction time) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Allan Wu, M.D., Principal Investigator — UCLA Neurology
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Siebner HR, Rossmeier C, Mentschel C, Peinemann A, Conrad B. Short-term motor improvement after sub-threshold 5-Hz repetitive transcranial magnetic stimulation of the primary motor hand area in Parkinson's disease. J Neurol Sci. 2000 Sep 15;178(2):91-4. doi: 10.1016/s0022-510x(00)00370-1. PMID 11018700
- [Background] Lang P. The international affective picture system [photographic slides]. Technical report. Gainsville, FL: The Center for Research in Phycophysiology, University of Florida; 1988.
- [Background] Tumas V, Rodrigues GG, Farias TL, Crippa JA. The accuracy of diagnosis of major depression in patients with Parkinson's disease: a comparative study among the UPDRS, the geriatric depression scale and the Beck depression inventory. Arq Neuropsiquiatr. 2008 Jun;66(2A):152-6. doi: 10.1590/s0004-282x2008000200002. PMID 18545773
- [Background] Filipovic SR, Rothwell JC, van de Warrenburg BP, Bhatia K. Repetitive transcranial magnetic stimulation for levodopa-induced dyskinesias in Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):246-53. doi: 10.1002/mds.22348. PMID 18951540
- [Background] Murase N, Rothwell JC, Kaji R, Urushihara R, Nakamura K, Murayama N, Igasaki T, Sakata-Igasaki M, Mima T, Ikeda A, Shibasaki H. Subthreshold low-frequency repetitive transcranial magnetic stimulation over the premotor cortex modulates writer's cramp. Brain. 2005 Jan;128(Pt 1):104-15. doi: 10.1093/brain/awh315. Epub 2004 Oct 13. PMID 15483042
- [Background] Lefaucheur JP, Fenelon G, Menard-Lefaucheur I, Wendling S, Nguyen JP. Low-frequency repetitive TMS of premotor cortex can reduce painful axial spasms in generalized secondary dystonia: a pilot study of three patients. Neurophysiol Clin. 2004 Oct;34(3-4):141-5. doi: 10.1016/j.neucli.2004.07.003. PMID 15501683
- [Background] Siebner HR, Mentschel C, Auer C, Conrad B. Repetitive transcranial magnetic stimulation has a beneficial effect on bradykinesia in Parkinson's disease. Neuroreport. 1999 Feb 25;10(3):589-94. doi: 10.1097/00001756-199902250-00027. PMID 10208595
- [Background] Khedr EM, Farweez HM, Islam H. Therapeutic effect of repetitive transcranial magnetic stimulation on motor function in Parkinson's disease patients. Eur J Neurol. 2003 Sep;10(5):567-72. doi: 10.1046/j.1468-1331.2003.00649.x. PMID 12940840
- [Background] Lefaucheur JP, Drouot X, Von Raison F, Menard-Lefaucheur I, Cesaro P, Nguyen JP. Improvement of motor performance and modulation of cortical excitability by repetitive transcranial magnetic stimulation of the motor cortex in Parkinson's disease. Clin Neurophysiol. 2004 Nov;115(11):2530-41. doi: 10.1016/j.clinph.2004.05.025. PMID 15465443
- [Background] Stern WM, Tormos JM, Press DZ, Pearlman C, Pascual-Leone A. Antidepressant effects of high and low frequency repetitive transcranial magnetic stimulation to the dorsolateral prefrontal cortex: a double-blind, randomized, placebo-controlled trial. J Neuropsychiatry Clin Neurosci. 2007 Spring;19(2):179-86. doi: 10.1176/jnp.2007.19.2.179. PMID 17431065
- [Background] Rektorova I, Sedlackova S, Telecka S, Hlubocky A, Rektor I. Dorsolateral prefrontal cortex: a possible target for modulating dyskinesias in Parkinson's disease by repetitive transcranial magnetic stimulation. Int J Biomed Imaging. 2008;2008:372125. doi: 10.1155/2008/372125. PMID 18274665
- [Background] Epstein CM, Evatt ML, Funk A, Girard-Siqueira L, Lupei N, Slaughter L, Athar S, Green J, McDonald W, DeLong MR. An open study of repetitive transcranial magnetic stimulation in treatment-resistant depression with Parkinson's disease. Clin Neurophysiol. 2007 Oct;118(10):2189-94. doi: 10.1016/j.clinph.2007.07.010. Epub 2007 Aug 21. PMID 17714987